CLINICAL TRIAL: NCT04106557
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Study to Evaluate the Efficacy and Safety of OV101 in Pediatric Individuals With Angelman Syndrome
Brief Title: A Study of OV101 in Individuals With Angelman Syndrome (AS)
Acronym: NEPTUNE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OV101-19-001
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Primary Disease or Condition Being Studied: Angelman Syndrome (AS)
MeSH Terms: interventions — gaboxadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant/Care Giver and Investigator/Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OV101 once daily (weight-based dosing) Other Name:Gaboxadol (Experimental): OV101 (gaboxadol), oral, provided once daily at bedtime for 12 week duration
  Interventions: Drug: Gaboxadol
- Placebo once daily (Placebo Comparator): Matching placebo,oral, provided once daily at bedtime for 12 week duration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gaboxadol — OV101 versus placebo once daily at bedtime for 12 weeks
  Arms: OV101 once daily (weight-based dosing) Other Name:Gaboxadol
Drug: Placebo — Matching placebo capsules to OV101 capsules.
  Arms: Placebo once daily

SUMMARY:
The purpose of this study is to assess the efficacy and safety of oral OV101 (gaboxadol) in pediatric subjects with Angelman syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and 2 to 12 years old (inclusive) at the time of informed consent
* Confirmed molecular diagnosis of AS
* Has a CGI-S-AS score of 3 or more at baseline.
* Meets the following age-appropriate body weight criterion:

  1. Subjects 2 to 3 years old must have a minimum body weight of 9 kg.
  2. Subjects 4 years and older must be between 17 kg and 64 kg (inclusive).
* Stable concomitant mediations for at least 4 weeks before study start

Exclusion Criteria:

* Any condition that would limit study participation
* Clinically significant lab or vital sign abnormalities at the time of screening
* Poorly controlled seizures (weekly seizures of any frequency with a duration more than 3 minutes, weekly seizures occurring more than 3 times per week, each with a duration of less than 3 minutes, or as defined by investigator assessment)
* Use of prescription medications for sleep, minocycline, or levodopa within the 4 weeks prior to Day 1 or during the study. Benzodiazepines chronically administered for seizure control are permitted.
* Cannot comply with protocol study assessments during screening or caregiver unable to comply with study requirements.
* Enrolled in any clinical trial or used any investigational agent within the 30 days before screening or concurrently with this study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (9):
  - Ovid Therapeutics Investigative Site, Phoenix, Arizona
  - Ovid Therapeutics Investigative Site, San Diego, California
  - Ovid Therapeutics Investigative Site, Chicago, Illinois
  - Ovid Therapeutics Investigative Site, Boston, Massachusetts
  - Ovid Therapeutics Investigative Site, Lexington, Massachusetts
  - Ovid Therapeutics Investigative Site, Cincinnati, Ohio
  - Ovid Therapeutics Investigative Site, Media, Pennsylvania
  - Ovid Therapeutics Investigative Site, Nashville, Tennessee
  - Ovid Therapeutics Investigative Site, Tacoma, Washington
- Australia (2):
  - Ovid Therapeutics Investigative Site, Brisbane, Queensland
  - Ovid Therapeutics Investigative Site, Heidelberg, Victoria
- Ovid Therapeutics Investigative Site, Munich, Germany
- Ovid Therapeutics Investigative Site, Ramat Gan, Israel
- Ovid Therapeutics Investigative Site, Rotterdam, Netherlands

REFERENCES:
- [Derived] Keary C, Bird LM, de Wit MC, Hatti S, Heimer G, Heussler H, Kolevzon A, Mathews A, Ochoa-Lubinoff C, Tan WH, Yan Y, Adams M. Gaboxadol in angelman syndrome: A double-blind, parallel-group, randomized placebo-controlled phase 3 study. Eur J Paediatr Neurol. 2023 Nov;47:6-12. doi: 10.1016/j.ejpn.2023.07.008. Epub 2023 Aug 1. PMID 37639777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Australia, Germany, Israel, and Netherlands.
Groups:
- OV101 Once Daily (Weight-based Dosing) Age 4 to 12: OV101 (gaboxadol), oral, provided once daily at bedtime for 12 week duration 4 to 12 years old
- OV101 Once Daily (Weight-based Dosing) Age 2 to 3: OV101 (gaboxadol), oral, provided once daily at bedtime for 12 week duration 2 to 3 years old
Period: Overall Study
Arm/Group | OV101 Once Daily (Weight-based Dosing) Age 4 to 12 | Placebo Once Daily | OV101 Once Daily (Weight-based Dosing) Age 2 to 3
Started | 47 | 50 | 7
Completed | 47 | 48 | 7
Not Completed | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- OV101 Once Daily (Weight-based Dosing) Age 4 to 12: OV101 (gaboxadol), oral, provided once daily at bedtime for 12 week duration
  Gaboxadol: OV101 versus placebo once daily at bedtime for 12 weeks
- OV101 Once Daily (Weight-based Dosing) Age 2 to 3: OV101 (gaboxadol), oral, provided once daily at bedtime for 12 week duration
- Total: Total of all reporting groups
Arm/Group | OV101 Once Daily (Weight-based Dosing) Age 4 to 12 | Placebo Once Daily | OV101 Once Daily (Weight-based Dosing) Age 2 to 3 | Total
Number analyzed (Participants) | 47 | 50 | 7 | 104
Age, Customized [Count of Participants; unit: Participants] — Population: Patients actual enroll
  Participants
    4-8 | 23 | 25 | 0 | 48
    9-12 | 24 | 25 | 0 | 49
    2-3 | 0 | 0 | 7 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 2 | 46
  Male | 23 | 30 | 5 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 0 | 7
  Not Hispanic or Latino | 44 | 46 | 7 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 1 | 0 | 4
  United States | 32 | 35 | 4 | 67
  Israel | 4 | 7 | 3 | 11
  Australia | 4 | 4 | 0 | 8
  Germany | 4 | 3 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impressions- Improvement in Angelman Syndrome (CGI-I-AS) Rating at 12 Weeks
Description: To evaluate the efficacy of OV101 versus placebo as assessed by the Clinical Global Impressions-Improvement-Angelman syndrome (CGI-I-AS) score at Week 12. CGIA-I-AS scores range from 1 (very much improved), to 4 (no change), to 7 (very much worse).
Time Frame: 12 weeks
Population: Total of 97 subjects, ages 4-12 years, inclusive. Participants aged 2 to 3 (n=7) did not participate in the scoring.
Measure: Count of Participants; unit: Participants
Groups:
- OV101 (Ages 4-12 Years, Inclusive): ages 4-12 years, inclusive taking OV101
- Placebo: ages 4-12 years, taking Placebo
Arm/Group | OV101 (Ages 4-12 Years, Inclusive) | Placebo
Number analyzed (Participants) | 47 | 50
Participants
  1-Very much improved | 1 | 2
  2-Much improved | 11 | 11
  3-Minimally improved | 11 | 11
  4-No change | 22 | 21
  5-Minimally worse | 1 | 5
  6-Much worse | 1 | 0
  7-Very much worse | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 Weeks
Groups:
- OV101 Once Daily (Weight-based Dosing) Other Name:Gaboxadol: OV101 (gaboxadol), oral, provided once daily at bedtime for 12 week duration
  Gaboxadol: OV101 versus placebo once daily at bedtime for 12 weeks Age (Actual) 4 to 12 Years at Screening
- OV101 Once Daily (Weight-based Dosing) Age 2-3: OV101 (gaboxadol), oral, provided once daily at bedtime for 12 week duration Age (Actual) 2 to 3 Years at Screening
Arm/Group | OV101 Once Daily (Weight-based Dosing) Other Name:Gaboxadol | Placebo Once Daily | OV101 Once Daily (Weight-based Dosing) Age 2-3
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/50 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/50 | 0/7
Other Adverse Events (participants affected / at risk) | 31/47 | 22/50 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OV101 Once Daily (Weight-based Dosing) Other Name:Gaboxadol (N=47) | Placebo Once Daily (N=50) | OV101 Once Daily (Weight-based Dosing) Age 2-3 (N=7)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OV101 Once Daily (Weight-based Dosing) Other Name:Gaboxadol (N=47) | Placebo Once Daily (N=50) | OV101 Once Daily (Weight-based Dosing) Age 2-3 (N=7)
Fatigue (General disorders) | 3 | 1 | 0
Generalized tonic-clonic seizure (General disorders) | 3 | 0 | 0
Irritability (General disorders) | 3 | 2 | 0
Somnolence (General disorders) | 3 | 0 | 1
Drooling (Nervous system disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1
URI (Infections and infestations) | 2 | 1 | 1
Contusion (Nervous system disorders) | 0 | 1 | 1
Ear Infection (Ear and labyrinth disorders) | 0 | 1 | 1
Insomnia (Nervous system disorders) | 1 | 2 | 1
Lethargy (Blood and lymphatic system disorders) | 0 | 1 | 1
Prolonged aPTT (Investigations) | 5 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 0
Seizure (Nervous system disorders) | 5 | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT04106557/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04106557/SAP_001.pdf